CLINICAL TRIAL: NCT03276546
Title: SHARE-D: a Decision Tool to Help Patients With, or at Risk of, Coronary Heart Disease Make Informed Lifestyle Choices: Feasibility Study
Brief Title: SHARE-D: a Decision Tool to Help Patients Make Informed Lifestyle Choices
Acronym: SHARE-D
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University, Belfast (Other)
Collaborators: Northern Ireland Chest Heart and Stroke (Other)
Responsible Party: Principal Investigator, Dr Margaret E Cupples, Professor, Queen's University, Belfast
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 16/LO/0655
Record Dates: First submitted 2017-08-31; First posted 2017-09-08 (Actual); Results first posted 2024-01-22 (Actual); Last update posted 2024-01-22 (Actual); Status verified 2024-01

CONDITIONS: Health Behavior
MeSH Terms: conditions — Health Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SHARE-D decision tool use (Experimental): The intervention, a shared decision-making tool ('SHARE-D'), which is a paper-based questionnaire, will be used jointly by a health professional and patient to facilitate decision-making about initiating change in physical activity or diet behaviour
  Interventions: Behavioral: shared decision-making tool (SHARE-D)

INTERVENTIONS:
Behavioral: shared decision-making tool (SHARE-D) — questionnaire
  Other Names: questionnaire

SUMMARY:
More information is needed about effective ways to help people begin to change their lifestyle behaviours, particularly physical activity and diet. The investigators propose to test a 'tool' that can be used to guide discussions between people and health professionals about their physical activity and diet habits, so that people may be supported better in making decisions about why and how they might begin to fit more exercise and healthy food into their daily routines and make long-term changes. The investigators will explore the feasibility of using this tool in general practice, reviewing behaviours after 1 and 3 months. Patients' and healthcare professionals' views of its use and how it influenced decisions will inform development of the tool's design and a study of its effectiveness in helping people to begin to change their behaviour and achieve healthy lifestyles.

DETAILED DESCRIPTION:
Healthier lifestyles, relating to physical activity and diet, reduce the risk of heart disease and stroke. However, making and sustaining lifestyle changes is difficult. More information is needed about effective ways to help people begin to change their lifestyle behaviours. The investigators propose to test the feasibility of using a 'tool' (the SHARED-D questionnaire) in guiding discussions between people and health professionals about physical activity and diet, and support people in making decisions about why and how they might begin to fit more exercise and healthy food into their daily routines. The 'tool' (SHARE-D) consists of questions to help people think about their personal circumstances and their motivation, opportunities, capabilities and priorities, and includes information about heart disease and stroke.

The investigators will explore the use of this tool in general practice, assessing patients' physical activity and diet behaviour after 1 and 3 months. Patients' and healthcare professionals' views of its use and how it influenced decisions will help to improve the tool's design. Participants' opinions regarding its format and method of delivery will inform future plans for its use and the design of a study of its effectiveness in helping people to begin to change their behaviour and achieve healthy lifestyles, hoping to lead to improved quality of life for people with heart disease and stroke.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 years or over
* With or at high risk of coronary heart disease
* Overweight or physically inactive

Exclusion Criteria:

* Unable to complete questionnaires
* Unable to make independent changes to physical activity or diet habits

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

RESULTS

PARTICIPANT FLOW:
Recruitment Details: recruited from general practice; July-October 2016
Groups:
- SHARE-D Decision Tool Use: The intervention, a shared decision-making tool ('SHARE-D'), which is a paper-based questionnaire, will be used jointly by a health professional and patient to facilitate decision-making about initiating change in physical activity or diet behaviour shared decision-making tool (SHARE-D): questionnaire
Period: Overall Study
Arm/Group | SHARE-D Decision Tool Use
Started | 23
Completed | 20
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | SHARE-D Decision Tool Use
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 15
  >=65 years | 8
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 13
Race (NIH/OMB) [Count of Participants; unit: Participants] — Number of participants in each race category
  Participants
    American Indian or Alaska Native | 0
    Asian | 0
    Native Hawaiian or Other Pacific Islander | 0
    Black or African American | 0
    White | 23
    More than one race | 0
    Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants] — Recruited from general practice, Northern Ireland, UK; data collected by questionnaire
  Participants
    United Kingdom | 23
BMI [Count of Participants; unit: Participants] — classification of participants based on categories of BMI
  Participants
    Normal (18.5 - 24.9 kg/m^2) | 1
    Overweight (25 - 29.9 kg/m^2) | 3
    Obese (30 - >40 kg/m^2) | 19
DINE (Fibre score) [Mean (Standard Deviation); unit: units on a scale] — DINE (Dietary Instrument for Nutritional Education) questionnaire data provide a numerical score for the fibre content of food consumed. The score is based on 19-item questionnaire related to the frequency of eating various foods for which fibre content has been analysed and a 'fibre' score attributed. Higher scores represent better outcomes/ healthier diet. A score <30 = low fibre intake; 30-40 = medium fibre intake; >40 = high fibre intake. Max score for fibre consumption is 88; minimum is 1.
  units on a scale | 35.35 (11.23)
DINE (unsaturated fat score) [Mean (Standard Deviation); unit: units on a scale] — The DINE (Dietary Instrument for Nutritional Education) questionnaire provides a numerical score for the unsaturated fat content of food consumed. The score is based on frequency of eating various foods for which unsaturated fat content has been analysed and an 'unsaturated fat' score attributed. Higher scores represent better outcomes/ healthier diet. A score <6 = unsaturated fat intake; 6-9 = medium unsaturated fat intake; >9 = high unsaturated fat intake. Minimum score is 3 ; maximum is 12.
  units on a scale | 5.91 (1.86)
Self-report of sedentary behaviour, based on number of hours/ day watching TV [Number; unit: number of participants] — Self-reported time (hours) spent in various activities during the week prior to completion of the Recent Physical Activity Questionnaire (RPAQ); measure of sedentary behaviour focused on numbers reporting watching TV for >2hrs/ weekday.
  number of participants | 14
Numbers doing >30minutes of MVPA/day (accelerometer data) [Count of Participants; unit: Participants] — accelerometer recording, measured over 7 days at baseline - objective measure of step counts and time spent (minutes/day) of sedentary behaviour and moderate and vigorous physical activity (MVPA); measure used in study to assess numbers doing >30minutes of MVPA/day (achieving physical activity recommendations)
  Participants | 6

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Rate
Description: numbers of patients attending a baseline assessment, compared to numbers invited to participate
Time Frame: 4 months overall recruitment (responses to invitations recorded within 4 weeks of invitation being sent)
Population: Responses recorded within 4 weeks of invitation being sent; participants enrolled were those who completed baseline assessment - recruitment constrained by availability of researcher, space in practice, other commitments of potential participants and study timeline
Measure: Count of Participants; unit: Participants
Groups:
- SHARE-D Decision Tool Use: The intervention, a shared decision-making tool ('SHARE-D'), which is a paper-based questionnaire, will be used jointly by a health professional and patient to facilitate decision-making about initiating change in physical activity or diet behaviour shared decision-making tool (SHARE-D): questionnaire
  Recruitment rate: 28% (45/162)
Arm/Group | SHARE-D Decision Tool Use
Number analyzed (Participants) | 162
Participants
  Number who responded positively to invitation | 45
  Number who attended baseline assessment | 23

2. Secondary Outcome: Completion Rate
Description: numbers of enrolled participants who complete all assessments and reviews
Time Frame: 3 months
Population: Number (%) of those who attended baseline assessments and completed all assessments and follow-up
Measure: Count of Participants; unit: Participants
Groups:
- SHARE-D Decision Tool Use: The intervention, a shared decision-making tool ('SHARE-D'), which is a paper-based questionnaire, will be used jointly by a health professional and patient to facilitate decision-making about initiating change in physical activity or diet behaviour shared decision-making tool (SHARE-D): questionnaire
  Recruitment rate: 28% (45/162); Completion rate 20/23 (87%)
Arm/Group | SHARE-D Decision Tool Use
Number analyzed (Participants) | 23
Participants | 20

3. Secondary Outcome: Diet Behaviour - Fibre Intake
Description: Dietary Instrument for Nutritional Education (DINE) questionnaire - measure of diet fibre content; maximum score = 61; minimum = 3; higher score indicates better outcome
Time Frame: 3 months
Population: Fibre score, higher score better diet
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | SHARE-D Decision Tool Use
Number analyzed (Participants) | 23
score on a scale
  Mean Fibre Score (SD) baseline | 35.35 (11.23)
  Mean Fibre Score (SD) 3 months: number analyzed (Participants) | 20
  Mean Fibre Score (SD) 3 months | 34.60 (11.81)

4. Secondary Outcome: Physical Activity Behaviour
Description: RPAQ questionnaire -self-reported frequency of episodes of different activities representing levels of sedentary behaviour and of light, moderate and vigorous physical activity in 4 weeks prior to completion of the questionnaire; focus on measure of sedentary behaviour indicated by time (hours) spent watching TV/weekday
Time Frame: 3 months
Population: Time spent watching TV>2hrs/weekday represents time spent in sedentary behaviour
Measure: Number; unit: participants
Arm/Group | SHARE-D Decision Tool Use
Number analyzed (Participants) | 23
participants
  Number watching TV>2hrs/weekday at baseline | 14
  Number watching TV >2hrs/ weekday at 3 months: number analyzed (Participants) | 20
  Number watching TV >2hrs/ weekday at 3 months | 16

5. Secondary Outcome: Objective Measure of Physical Activity
Description: accelerometer measurement of duration of light, moderate and vigorous physical activity per day over a 7-day period
Time Frame: 2 periods of 7-day measurement: baseline and after 3 months
Population: accelerometer measurement of duration of moderate and vigorous physical activity (MVPA) per day over a 7-day period, measuring number achieving 30 minutes of MVPA/day at baseline and after 3 months
Measure: Count of Participants; unit: Participants
Arm/Group | SHARE-D Decision Tool Use
Number analyzed (Participants) | 23
Participants
  achieved 30 mins MVPA/day at baseline | 16
  achieved 30 mins MVPA/day at 3 months | 5
  did <30 mins MVPA/day at baseline | 10
  did <30mins/day MVPA at 3 months | 11

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | SHARE-D Decision Tool Use
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-07): https://cdn.clinicaltrials.gov/large-docs/46/NCT03276546/Prot_SAP_000.pdf